CLINICAL TRIAL: NCT07140848
Title: A Novel Continuous Glucose Monitoring Enhanced DPP Intervention to Prevent Type 2 Diabetes in Adults With Prediabetes
Brief Title: CGM-Enhanced DPP to Prevent Type 2 Diabetes in Adults With Prediabetes
Acronym: CGM-DPP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Raphael Fraser, PhD, Associate Professor of Medicine, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00009767; ADA Grant #7-25-ICTSPC-412 (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2025-08-22; First posted 2025-08-26 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: PreDiabetes
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Active Comparator): Diabetes Prevention Program
  Interventions: Behavioral: Control
- Intervention (Experimental): Diabetes Prevention Program + Continuous Glucose Monitors/Coaching
  Interventions: Behavioral: CGM-DPP

INTERVENTIONS:
Behavioral: CGM-DPP — Participants in the DPP who receive personalized CGM coaching.
  Arms: Intervention
Behavioral: Control — Participants in control group will be referred to DPP.
  Arms: Control

SUMMARY:
Prediabetes affects over one-third of adults in the United States, placing them at a higher risk for developing type 2 diabetes and heart disease, which can lead to serious health complications and increased medical costs. Although a program called the Diabetes Prevention Program (DPP) has been shown to lower the risk of diabetes through healthy lifestyle changes, many people find it difficult to stick with these changes over the long term. This study seeks to find out if combining DPP coaching with continuous glucose monitoring (CGM) technology can help people stay on track with their health goals.

DETAILED DESCRIPTION:
CGM devices give individuals real-time information about their blood sugar levels, which can help them understand how their diet, exercise, and daily habits impact their health. By pairing CGM technology with support from trained DPP coaches, this approach aims to make it easier for participants to maintain healthy behaviors. The study will involve 214 adults with prediabetes who will follow a 12-month program with regular check-ins to measure improvements in blood sugar control, weight loss, physical activity, and overall quality of life.

The goal is to show whether using CGM in combination with coaching can lead to better health outcomes and whether it is a cost-effective way to prevent diabetes. If successful, this approach could be used in healthcare settings across the country, helping more people prevent diabetes and lead healthier lives.

ELIGIBILITY:
Inclusion Criteria:

1. adults aged 18 years or older,
2. diagnosis of prediabetes, as defined by current clinical guidelines (HbA1c 5.7% to 6.4%, fasting plasma glucose 100-125 mg/dL, or 2-hour plasma glucose 140-199 mg/dL following a 75g oral glucose tolerance test),
3. body mass index (BMI) of at least 24 kg/m² (or 22 kg/m² for Asian Americans),
4. willingness to comply with all aspects of the study protocol, including attending coaching sessions and using CGM devices.

Exclusion Criteria:

Individuals will be excluded from the study if they

1. have a diagnosis of type 1 or type 2 diabetes,
2. are currently using CGMs or have medical contraindications to CGM use, such as severe skin allergies or implantable defibrillators, or
3. are currently enrolled in another clinical trial for prediabetes. Additionally, using validated assessments, we will exclude participants with significant dementia, alcohol or drug abuse/dependency, active psychosis, or life expectancy less than 12 months as these conditions are likely to interfere with adherence to the intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2028-01-02 (Estimated); Study Completion 2028-01-02 (Estimated)

PRIMARY OUTCOMES:
Glycemic Control (HbA1c) | Change from baseline HbA1c at 12 months post intervention follow-ups
  Blood specimens (10 cc of blood) will be obtain by trained phlebotomists or nurse for HbA1c.

SECONDARY OUTCOMES:
Quality of Life as measured by SF-12 | Change from baseline quality of life measure at 12 months post intervention follow-ups
  The SF-12 (Ware 1996) is a valid and reliable instrument to measure functional status and reproduces 90% of the variance in PCS-36 and MCS-36 scores.

OTHER OUTCOMES:
Self-Care | Change from baseline self-care at 12 months post intervention follow-ups
  Behavioral skills will be assessed with the Summary of Diabetes Self-Care Activities (SDSCA) scale (Toobert 2000), a brief, validated questionnaire of diabetes self-care.